CLINICAL TRIAL: NCT04939090
Title: A Randomized Phase III Trial of Olanzapine Versus Megestrol Acetate for Cancer-Associated Anorexia
Brief Title: Olanzapine Versus Megestrol Acetate for the Treatment of Loss of Appetite Among Advanced Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A222004; NCI-2021-03303 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH)
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Advanced Malignant Solid Neoplasm; Anorexia; Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Anorexia; Hematologic Neoplasms | interventions — Olanzapine; Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (olanzapine) (Experimental): Patients receive olanzapine PO QD for up to 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olanzapine; Other: Questionnaire Administration
- Arm II (megestrol acetate) (Active Comparator): Patients receive megestrol acetate PO QD for up to 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Megestrol Acetate; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Olanzapine — Given PO
  Arms: Arm I (olanzapine)
Drug: Megestrol Acetate — Given PO
  Arms: Arm II (megestrol acetate)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares the effects of olanzapine versus megestrol acetate in treating loss of appetite in patients with cancer that has spread to other places in the body (advanced). Olanzapine may stimulate and increase appetite. This study aims to find out if olanzapine is better than the usual approach (megestrol acetate) for stimulating appetite and preventing weight loss.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVE:

I. To determine whether olanzapine leads to greater appetite improvement from baseline in cancer patients suffering from anorexia compared to megestrol acetate using the 0-10 numerical rating scale (NRS).

SECONDARY OBJECTIVES:

I. To determine whether olanzapine leads to a greater proportion of patients who report a 5% or greater weight gain from baseline compared to megestrol acetate.

II. To compare change in cachexia/anorexia symptoms with olanzapine compared to megestrol acetate using the Functional Assessment of Anorexia/Cachexia Treatment (FAACT)-Anorexia/Cachexia Subscale (A/CS) instrument.

OUTLINE: Patient are randomized to 1 of 2 arms.

ARM I: Patients receive olanzapine orally (PO) once daily (QD) for up to 4 weeks in the absence of consent withdrawal or unacceptable toxicity.

ARM II: Patients receive megestrol acetate PO QD for up to 4 weeks in the absence of consent withdrawal or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study due to the teratogenic potential of the therapy utilized in this trial. Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives or double barrier method (diaphragm plus condom)
* Diagnosis of advanced cancer
* Patient-reported 2-month weight loss of at least 5 pounds (2.3 kilograms) and/or physician-estimated caloric intake of less than 20 calories/kilogram of body weight per day
* The patient must perceive loss of appetite and/or weight as a problem; and have an appetite score of 4 or worse on the "Please rate your appetite…." question that requires a patient response on a 0-10 numeric rating scale
* Not receiving ongoing tube feedings or parenteral nutrition at the time of registration
* Not currently using systemic adrenal steroids (with the exception of short-term dexamethasone within 3 days of chemotherapy for control of chemotherapy side effects)
* No use of androgens, progesterone analogs, or other appetite stimulants within the past month
* Patient should not have poorly controlled hypertension or congestive heart failure at registration
* Patient should not have an obstruction of the alimentary canal, malabsorption, or intractable vomiting (defined as vomiting more than 3 times per day over the preceding week)
* Not currently using olanzapine for another medical condition or had previously used olanzapine for chronic nausea or for any pre-existing psychotic disorder
* Patient should not have had a previous blood clot at any time in the past
* No history of poorly controlled diabetes
* No symptomatic leptomeningeal disease or known brain metastases as these patients may have difficulty taking oral medications
* No history of hypersensitivity to olanzapine or megestrol acetate
* No COVID-19 infection in the past that, in the opinion of the treating physician, had left patients with compromised taste, which has not resolved at the time of registration
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential only, a negative urine or serum pregnancy test done =< 14 days prior to registration is required
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Estimated life expectancy of 3 months or longer
* Serum creatinine =< 2.0 mg/dL
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 3 x upper limit of normal (ULN)
* Fasting glucose < 140 mg/dL
* Granulocytes > 1000/hpf
* No treatment with another antipsychotic agent, such as risperidone, quetiapine, clozapine, butyrophenone within 30 days of enrollment
* In order to complete the mandatory patient-completed measures, participants must be able to speak and/or read English or Spanish. Sites seeking to enroll Spanish-speaking patients should have access to Spanish speaking staff on site or through the use of a translation service to be able to conduct the informed consent discussion in Spanish, and to conduct the weekly phone calls

Exclusion Criteria:

* Psychiatric illness which would prevent the patient from giving informed consent
* Medical condition such as uncontrolled infection (including human immunodeficiency virus [HIV]), uncontrolled diabetes mellitus or cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
* Patients who cannot swallow oral formulations of the agents
* Patients with impaired decision-making capacity (such as with a diagnosis of dementia or memory loss) are not eligible for this study
* No presence of a hormone-sensitive tumor, such as breast, endometrial, or prostate cancer (this exclusion criterion is intended to circumvent any confounding antineoplastic effects of megestrol acetate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in appetite | Baseline up to 4 weeks
  Will be compared between the two study groups (olanzapine versus megestrol acetate) using a 0-10 numerical rating scale. Will be summarized by mean (standard deviation [SD]) and median (range) by treatment arm. The difference in appetite change from baseline to 4 weeks of treatment between arms will be estimated along with a 95% confidence interval and will be compared using a t-test or Wilcoxon rank-sum test as appropriate.

SECONDARY OUTCOMES:
Proportion of patients who report a 5% or greater weight gain | Baseline up to 4 weeks
  The proportion of patients with a 5% or greater weight gain from baseline will be calculated for each arm. The difference in proportion of patients with 5% or greater weight gain between the arms will be estimated along with a 95% confidence interval using a normal approximation of the binomial distribution and will be compared using a Chi-squared test.
Change in well-being status and cachexia/anorexia symptoms | Baseline up to 4 weeks
  Responses to the Functional Assessment of Anorexia/Cachexia Treatment (FAACT)-Anorexia/Cachexia Subscale (A/CS) questionnaire will be scored according to the established algorithm. The total score of the FAACT-A/CS will be summarized weekly and the change from baseline to 4 weeks will be compared between the treatment arms using the same methods described for the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (293):
- United States (293):
  - Arizona Center for Cancer Care - Gilbert, Gilbert, Arizona
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Arizona Center for Cancer Care - Phoenix, Phoenix, Arizona
  - Arizona Center for Cancer Care - Osborn, Scottsdale, Arizona
  - Arizona Center for Cancer Care - Scottsdale, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Epic Care-Dublin, Dublin, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Washington Hospital, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Bay Area Tumor Institute, Oakland, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - Dominican Santa Cruz Hospital, Santa Cruz, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Halifax Health Center for Oncology - Ormond Beach, Ormond Beach, Florida
  - South Florida Baptist Hospital, Plant City, Florida
  - Halifax Health Center for Oncology - Port Orange, Port Orange, Florida
  - Mease Countryside Hospital, Safety Harbor, Florida
  - Saint Anthony's Hospital Cancer Care Center, St. Petersburg, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Piedmont Newnan Hospital, Newnan, Georgia
  - Piedmont Henry Hospital, Stockbridge, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente Lutherville - Timonium Medical Center, Lutherville, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Exeter Hospital, Exeter, New Hampshire
  - Hunterdon Medical Center, Flemington, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Glens Falls Hospital, Glens Falls, New York
  - Queens Hospital Center, Jamaica, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Levine Cancer Institute - Rutherford, Forest City, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Regional Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Baptist Hospitals of Southeast Texas Cancer Center, Beaumont, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Tarrant County Hospital District/JPS Health Network, Fort Worth, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Kaiser Permanente-Caton Hill Medical Center, Woodbridge, Virginia
  - Valley Medical Center, Renton, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes